CLINICAL TRIAL: NCT04464642
Title: Tofacitinib Versus Methotrexate as the First Line DMARD in the Treatment of Rheumatoid Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. Mohammad Mamun Khan (Other)
Responsible Party: Sponsor-Investigator, Dr. Mohammad Mamun Khan, Resident, BSMMU, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Organization: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU /2019/5499
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis tofacitinib methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; tofacitinib

STUDY DESIGN:
Intervention Model Description: open label Randomization controlled clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): group "A" is a control arm who will get conventional drug (methotrexate). 25 mg subcutaneous weekly . at 3 months if DAS-28 not fall by at least 1.2, drug is to be changed and regarded as therapy failure. if at least 1.2 improvement of DAS-28 occur,then therapy is continued for 6 monyhs
  Interventions: Drug: Methotrexate
- group B (Experimental): group "B" will get tofacitinib 10 mg weekly. if DAS-28 not improved at least 1.2 at 3 months, it is regarded as therapy failure. if improved at least 1.2, then therapy continued for 6 months
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 25 mg subcutaneous is given in group A
  Other Names: injection trexonate
  Arms: group A
Drug: Tofacitinib — tofacitinib 10 mg given in group B
  Other Names: tofacit
  Arms: group B

SUMMARY:
It is a randomized controlled study

DETAILED DESCRIPTION:
Randomization controlled study on Rheumatoid arthritis patients whos disease activity is high, controlled subjects will be given methotrexate and study subjects will get tofacitinib

ELIGIBILITY:
Inclusion Criteria:1. age greater than 18 years 2. patients fulfill the ACR-EULAR classification criteria for RA 3.DAS-28 CRP more than 5.1

-

Exclusion Criteria:

1. systemic infection
2. hemoglobin less than 9 mg/dl
3. WBC <4000, neutrophil <1000, platelet <100000/mm
4. live vaccine within 3 months
5. GFR < 50 ml/min
6. ALT > 2 times ULN
7. pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
DAS-28 CRP at 6 month | 6 months
  disease activity score in 28 joints has to measured at 6 months

SECONDARY OUTCOMES:
SDAI at 6 months | 6 months
  simplified disease activity index at 6 months
HAQ-DI at 6 months | 6 months
  health assesment by HAQ-DI at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad M Khan, MBBS, Principal Investigator — Resident doctor, BSMMU
Locations (1):
- Bangabandhu Seikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan MM, Ahmed S, Hasan Sajib MK, Morshed AA, Mahbub-Uz-Zaman K, Haq SA. Tofacitinib versus methotrexate as the first-line disease-modifying antirheumatic drugs in the treatment of rheumatoid arthritis: An open-label randomized controlled trial. Int J Rheum Dis. 2023 Sep;26(9):1729-1736. doi: 10.1111/1756-185X.14801. Epub 2023 Jun 28. PMID 37377385